CLINICAL TRIAL: NCT04434014
Title: Proper Nutrition and Its Relationship to Oral Diseases in the Era of Corona
Brief Title: Proper Nutrition And Its Relation To Oral Diseases In Covid -19 Era
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Samah Mohamed Kamel, associate professr, October University for Modern Sciences and Arts
Other Study IDs: 12345678
Record Dates: First submitted 2020-06-06; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Diet, Healthy
Keywords: Proper Diet; Taste; Oral Health; Corona

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- males from 20 to above 65 y: will be sub divided into 4 groups according to age sub group I from 20 - 35 sub group II from 36- 45 sub group III from 46- 65 sub group IV more than 65
  Interventions: Dietary Supplement: proper diet
- female from 20 to above 65 y: will be sub divided into 4 groups according to age will be sub divided into 4 groups according to age sub group I from 20 - 35 sub group II from 36- 45 sub group III from 46- 65 sub group IV more than 65
  Interventions: Dietary Supplement: proper diet

INTERVENTIONS:
Dietary Supplement: proper diet — diet containing all essential vitamins

SUMMARY:
effect of proper diet and vitamins on the oral health and the regeneration of the taste and smell in Covid 19 patients

DETAILED DESCRIPTION:
effect of proper diet and vitamins on the oral health ( bleeding gums, ulcers, bad breath) also the effect of proper diet on the regeneration of the taste and smell in Covid 19 patients A diet will be followed for 2 weeks then the progress will be evaluated by making another questionnaire

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* chronic diseases

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: * the participants will answer a questionnaire then a diet will be sent to the participants
  * the participants will follow the sent diet for 2 weeks then another questionnaire will be sent to the participants
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-06-18 (Estimated); Study Completion 2020-06-28 (Estimated)

PRIMARY OUTCOMES:
regeneration of taste | 2 weeks
  counting the fungiform papillae in 1cm x 1cm area of the tongue during the infection and after being cured

CONTACTS AND LOCATIONS:
Locations (1):
- October university of modern sciences and arts, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No